CLINICAL TRIAL: NCT07078123
Title: Risk of Hydrocelectomy After Laparoscopic Living Donor Nephrectomy
Brief Title: Hydrocelectomies in Male Donors
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Amit Garg, Nephrologist, Professor or Medicine, Epidemiology and Biostatistics, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: REB25-0054
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hydrocele; Hydrocele of Tunica Vaginalis; Hydrocelectomy; Living Kidney Donor; Living Kidney Donation; Laparoscopic Nephrectomy
Keywords: hydrocele; living kidney donor; hydrocelectomy; laparoscopic nephrectomy
MeSH Terms: conditions — Testicular Hydrocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male Living Kidney Donors: Male kidney donors who had a laparoscopic nephrectomy between April 1, 2002 and March 31, 2020, at transplant centres in the province of Alberta, Canada. Each donor's nephrectomy date will serve as their cohort entry date.
  Interventions: Procedure: Laparoscopic Donor Nephrectomy
- Male Non-Donors: A similarly healthy segment of the general Alberta population selected using restriction and matching to emulate the health criteria required to be met for living kidney donation. We will randomly assign a cohort-entry date (simulated nephrectomy date) to all male residents in Alberta, according to the distribution of cohort-entry dates among donors (between April 1, 2002 and March 31, 2020).

INTERVENTIONS:
Procedure: Laparoscopic Donor Nephrectomy — Receipt of a laparoscopic nephrectomy for kidney donation
  Groups: Male Living Kidney Donors

SUMMARY:
This is a population-based matched cohort study to examine whether male living kidney donors are at increased risk of undergoing hydrocelectomy compared to similar males in the general population. Using linked health administrative data from Alberta, Canada, male donors who underwent laparoscopic nephrectomy between 2002 and 2020 will be matched 1:10 to non-donors based on key demographic and clinical characteristics. Males will be followed for several years, from the time of cohort entry through the datasets until March 2021. The primary outcome is a hospital admission for hydrocelectomy in the follow-up period. The secondary outcome is receipt of a scrotal ultrasound.

DETAILED DESCRIPTION:
*Summary*

Background: Some male living kidney donors experience scrotal pain and swelling on the same side as their nephrectomy following donation, occasionally requiring surgical intervention for relief.

Methods: In a population-based cohort study, we will identify male living kidney donors who underwent laparoscopic nephrectomy in Alberta, Canada, between 2002 and 2020. Each donor will be matched 1:10 to male non-donors from the general Alberta population with similar baseline health characteristics. Matching variables will include age, cohort entry date, rural versus urban residence, income quintile, prior vasectomy, and history of inguinal hernia repair. Donors and non-donors will be followed using linked provincial healthcare administrative databases in Alberta, Canada, until March 31, 2021. The primary outcome will be hospital admission for hydrocelectomy. The secondary outcome will be the receipt of a scrotal ultrasound.

Study Objective: This study aims to determine whether male living kidney donors who undergo laparoscopic nephrectomy have a higher risk of hydrocelectomy compared to matched male non-donors with similar baseline health profiles.

*Background*

Understanding the risks associated with living kidney donation is essential for ensuring informed consent, guiding donor follow-up, and identifying potential opportunities to reduce harm. While most donors recover well, emerging evidence suggests that some male donors may experience postoperative scrotal pain and swelling on the side of their nephrectomy. In this years following donation, these symptoms can lead to surgical intervention such as hydrocelectomy.

*Study Design and Setting*

We propose a population-based matched cohort study using linked administrative health data from the Alberta Kidney Disease Network (AKDN), which includes datasets from Alberta Health, the provincial health ministry. Over 99% of Alberta residents are registered for provincial health coverage, ensuring near-complete population capture of hospital care and physician services.

We are publishing the study protocol a priori to conducting statistical analyses including outcome analyses to strengthen methodological rigour and transparency. This study adheres to the STROBE and RECORD reporting guidelines and has received research ethics approval from the Universities of Alberta and Calgary, with a waiver of informed consent due to the use of de-identified administrative data.

*Data Sources*

Baseline characteristics and outcomes are derived from AKDN-linked datasets, including physician claims, hospital discharge abstracts, provincial laboratory data, and pharmacy records. Alberta adopted the Canadian Classification of Health Interventions (CCI) in April 2002, which defines the start of the accrual period. Laboratory data includes serum creatinine and urine albumin from 2002 onward. These databases have been validated and widely used in prior health services research.

*Study Population*

We will include all male Alberta residents who underwent living donor nephrectomy between April 1, 2002, and March 31, 2020. Donors will be identified using the algorithm of an ICD-10 code for kidney donation (Z52.4) and a CCI procedural code for kidney procurement or excision (1.PC.58, 1.PC.89, or 1.PC.91). The date of donation nephrectomy will be the index date. Donors will be excluded if they are under 18, out-of-province, have incomplete demographic data, died on or before the nephrectomy date, or had prior dialysis, organ transplant, or scrotal procedures (excluding vasectomy or inguinal hernia repair), scrotal ultrasound. For the primary analysis we will concentrate on males who had a laparoscopic donor nephrectomy and exclude those who underwent an open donor nephrectomy, as in prior studies scrotal complications more prevalent after laparoscopic nephrectomy compared to open nephrectomy.

The non-donor comparator group will be drawn from the general population of all adult males in Alberta. Among this cohort, we will exclude those with comorbidities that would contraindicate donation, those without at least one physician visit in the previous two years, and those with prior scrotal conditions. The non-donor index date will be randomly assigned to all males in Alberta based on the distribution of the donors' nephrectomy dates (2002-2020). Each donor will be matched to 10 non-donors based on age (±1 year), cohort entry year (±3 years), rural/urban residence, income quintile, prior vasectomy, and prior inguinal hernia repair.

*Baseline Characteristics*

Baseline variables will be assessed at the index date (i.e. the nephrectomy date in the donor group or simulated index date for non-donors). Demographic data (age, sex, rurality, income quintile) will be obtained from Alberta Health records and census files. Clinical characteristics such as comorbidities, estimated glomerular filtration rate (eGFR), and albuminuria will be obtained from hospital discharge records, outpatient laboratory data, and physician claims data preceding the index date.

*Outcomes*

Participant observation time will be censored at the time of death, emigration, or until the maximum follow-up date (March 31, 2021). The primary outcome is a hospital admission for hydrocelectomy confirmed through both a receipt of a physician billing code (AHCIP: 73.0, 73.0A, 73.1, 73.1A, 73.1B, 73.9, 73.91, 75.0) and a hospital procedural code (CCI: 1QH87LA, 1QH87LB, 1QH52HA, 1QH52LA, 1QH80LA, 1QG52HA, 1QG52LA) within 30 days of one another. The secondary outcome will be the receipt of a scrotal ultrasound. Data on laterality of the nephrectomy is not available, but ~90% of donor nephrectomies are expected to be left-sided. Data on the laterality of the hydrocelectomy is not available.

*Statistical Analysis Plan*

Baseline characteristics will be compared using standardized mean differences, with >10% indicating a meaningful difference. We will use Cox proportional hazards models with robust variance estimation to account for matched sets and estimate hazard ratios for our outcomes. Proportional hazards assumptions will be evaluated using Kolmogorov-type supremum tests; if violated, stratified log-rank tests and differences in 20-year restricted mean survival time will be used. Outcomes will be described as incidence rates per 1000 person-years and cumulative incidence. These results will be obtained using the Aalen-Johansen estimator, counting the first event and treating death as a competing event, where donors and nondonors will be compared visually with graphical curves and at prespecified time points.

Prespecified secondary analyses will include a comparison of donors who underwent laparoscopic versus open nephrectomy. Inverse probability of treatment weighting (IPTW) from propensity scores will be used to balance covariates across the groups. All statistical tests will be two-sided, using a hierarchical testing framework. We will use R version 4.2.3 to conduct analyses, with significance defined as p < 0.05.

* P values (significance testing) and confidence intervals *: We will perform hierarchical statistical tests to assess our hypotheses in the pre-defined order described below. The 2-sided significance level will be 0.05 for each tested hypothesis. After a non-significant test no further significance testing will be performed and no further P values will be reported. All estimates (with and without P values) will be reported as point estimates with 95% confidence intervals. We acknowledge the interval widths of the estimates without P values are not adjusted for multiple testing and that those inferences may not be reproducible. The order:

(i) the primary outcome (hydrocele surgery) in donors vs. nondonors (ii) the secondary outcome (scrotal ultrasound) in donors vs. nondonors (iii) primary outcome in donors who underwent a laparoscopic vs. open procedure (iv) secondary outcome in donors who underwent a laparoscopic vs. open procedure.

ELIGIBILITY:
Donors: We will include male individuals who underwent laparoscopic donor nephrectomy in Alberta, Canada, between April 1, 2002, and March 31, 2020.

* Individuals with data record errors (e.g., missing or invalid age, sex, or date of birth), who are less than 18 years of age or greater than 105 years of age, who have a death record on or before the date of nephrectomy, or have a date of last contact <4 months after cohort entry (i.e., they don't live permanently in the province), will be excluded.
* Those with evidence of prior dialysis or a previous solid organ transplant will be excluded.
* Individuals who have no physician visits within the last year will be excluded.
* Individuals who, prior to donation, underwent a scrotal ultrasound or a scrotal procedure, other than a vasectomy or inguinal hernia repair, will be excluded.
* We will exclude those who had an open nephrectomy, focusing on those who underwent laparoscopic surgery.

Non-donors: Before nephrectomy, living donors undergo rigorous health screening, thus. we will select a similarly healthy cohort of the general population using restriction and matching. We will randomly assign a cohort-entry date (simulated nephrectomy date) to all male persons who were citizens in Alberta, according to the distribution of cohort-entry dates among donors (April 1, 2002, to March 31, 2020). To emulate the health status of living donors, we will further restrict the sample to exclude individuals with medical conditions that would typically preclude donation.

Using data prior and at the time of cohort entry we will exclude:

* Individuals with data record errors (e.g., missing or invalid age, sex, or date of birth), who are less than 18 years of age or greater than 105 years of age, with a death record on or before their cohort entry, or have a date of last contact <4 months after cohort entry (to restrict to permanent residents of the province)
* Those with evidence of prior dialysis or a previous solid organ transplant.
* Any hospitalization for mental illness, palliative care, or multiple admissions in the prior year and any admission to an intensive care unit in the prior year.
* High comorbidity, based on the Charlson comorbidity index (≥3) in the last 5 years.
* Any resident in a long-term care facility or diagnosed with dementia.
* Any history of kidney disease (including nephrology consultation, kidney biopsy, acute kidney disease, chronic kidney disease, or any disorders of the kidneys, ureters or bladder).
* Any history of cardiovascular disease (including congestive heart failure, myocardial infarction, peripheral vascular disease, ischemic stroke, abdominal aortic aneurysm repair, or hypertension in individuals under 50 years of age).
* Any form of cancer in the last five years, any history of liver disease or cirrhosis, diabetes, or serious infections such as hepatitis, HIV, or infective endocarditis.
* Any autoimmune rheumatic conditions (including rheumatoid arthritis and systemic lupus erythematosus).
* Any documented history of alcoholism in the last 5 years.
* More than four family physician visits in the past two years (which suggests they have active medical issues).
* No family physician visits in the past two years (to ensure they have access to a primary care physician).
* Individuals who, prior to their assigned cohort entry date, underwent a scrotal ultrasound or a scrotal procedure, other than a vasectomy or inguinal hernia repair.

Matching

Donors will be matched 1:10 to eligible non-donors based on baseline characteristics that may influence the risk of undergoing a hydrocelectomy. Matching criteria will include:

* Age at cohort entry, as the risk of hydrocele increases with age in adult males.
* Cohort entry year, to account for potential temporal or era effects.
* Urban vs. rural residence (defined by population ≥10,000 vs. <10,000), given that rural residence may be associated with reduced access to care and poorer health outcomes.
* Neighbourhood income quintile, as individuals from lower-income areas may face barriers to healthcare access and experience worse outcomes.
* History of vasectomy and history of inguinal hernia repair, as both procedures can sometimes result in chronic testicular pain, which may be related to later hydrocelectomy.

Each non-donor will be matched to only one donor, without replacement.

Ages: 18 Years to 106 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will include all male Alberta residents who underwent living donor nephrectomy between April 1, 2002, and March 31, 2020. The date of donation nephrectomy will be the index date. The non-donor comparator group will be drawn from the general population of all adult males in Alberta. The non-donor index date will be randomly assigned to all males in Alberta based on the distribution of the donors' nephrectomy dates (2002-2020). Each donor will be matched to 10 non-donors.
Sampling Method: Non-Probability Sample
Enrollment: 2750 (Estimated)
Dates: Start 2002-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Hydrocelectomy | Donors and their matched non-donors will enter the cohort between April 1, 2002 and March 31, 2020, and will be followed until study outcome (first event), death, emigration from the province, or the end of the observation period (March 31, 2021).
  Hospital admission and receipt of surgery for a hydrocele excision. To be confident in outcome ascertainment, evidence of both a surgeon-fee-for-service code and a hospital-based procedural code will be required, with each recorded in separate healthcare databases by different personnel.
  1 AHCIP code and 1 CCI code within 30 days: CCI: 1QH87LA, 1QH87LB, 1QH52HA, 1QH52LA, 1QH80LA, 1QG52HA, 1QG52LA AHCIP: 73.0, 73.0A, 73.1, 73.1A, 73.1B, 73.9, 73.91, 75.0

SECONDARY OUTCOMES:
Scrotal Ultrasound | Donors and their matched non-donors will enter the cohort between April 1, 2002 and March 31, 2020, and will be followed until study outcome (first event), death, emigration from the province, or the end of the observation period (March 31, 2021).
  Receipt of a scrotal ultrasound. This test is typically ordered to evaluate a person with ongoing pain or swelling in their scrotum or testis.
  CCI: 3.QG.30 AHCIP: X330

IPD SHARING:
Plan to Share IPD: No
The dataset from this study is held securely in coded form with an Alberta Kidney Disease Network Analyst. Provincial privacy regulations prohibit making the dataset publicly available.